CLINICAL TRIAL: NCT03931759
Title: The Effect of Intra-abdominal Pressure, Applied to the Patients Diagnosed With Diabetes Mellitus, Who Undergo Laparoscopic Surgery, on Hemodynamics
Brief Title: The Effect of Intra-abdominal Pressure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, Nurhan EREN, research assistant, Erzincan University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: EBYU1
Record Dates: First submitted 2019-04-23; First posted 2019-04-30 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Diabetes Mellitus; ASA Triad; Cardiac Autonomic Neuropathy
Keywords: diabetes mellitus; cardiac autonomic neuropathy; laparoscopic surgery
MeSH Terms: conditions — Diabetes Mellitus; Asthma, Nasal Polyps, And Aspirin Intolerance | interventions — Laparoscopy

STUDY DESIGN:
Intervention Model Description: prospective randomize clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diabetes mellitus (Active Comparator): patients with diabetes mellitus
  Interventions: Diagnostic Test: laparoscopic surgery
- non-Diabetes mellitus (No Intervention): patients without diabetes mellitus

INTERVENTIONS:
Diagnostic Test: laparoscopic surgery — patients with diabetes mellitus in laparoscopic surgery
  Other Names: hearth rate variability
  Arms: Diabetes mellitus

SUMMARY:
The Effect of Intra-abdominal Pressure

DETAILED DESCRIPTION:
The Effect of Intra-abdominal Pressure, Applied to the Patients Diagnosed with Diabetes Mellitus, Who Undergo Laparoscopic Surgery, on Hemodynamics

ELIGIBILITY:
Inclusion Criteria:

* diabetes mellitus
* laparoscopic surgery

Exclusion Criteria:

* hypertension
* hearth failure
* renal failure
* hepatic failure
* difficult intubation
* shock

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
The measurement of heart rate variability in laparoscopic surgeries | 1 year
  The measurement of heart rate variability is used as a method to assess the autonomic nerve system. As the autonomic nerve system dysfunction may complicate the possible peroperative problems in the patients to be operated, the pre-assessment of the autonomic nerve system function should be considered as an acquisition required to be obtained in the daily anesthesia practice.
  When we increase the intraabdominal pressure during the laparoscopic surgery, we think that the hemodynamic responses of the diabetic patient group, especially the patients with autonomic neuropathy, to this increasing intraabdominal pressure will be different. The aim of the present study is to investigate the effect of the intraabdominal pressure, applied to the patients diagnosed with diabetes mellitus who will have laparoscopic surgery, on hemodynamics.

IPD SHARING:
Plan to Share IPD: No